CLINICAL TRIAL: NCT01033695
Title: Interobserver Agreement of Endoscopic Ultrasonography and Endoscopic Sonoelastography in the Evaluation of Lymph Nodes
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Michael Bau Mortensen, Centre of Surgical Ultrasound
Other Study IDs: 12-2009
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-08

CONDITIONS: Lymph Nodes; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Liver Cancer
Keywords: Endoscopy; Endoscopic Ultrasound; Endoscopic Sonoelastography; Cancer; Interobserver agreement
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Endoscopic ultrasound (EUS) is an important part of the pre-treatment evaluation of patients with upper gastrointestinal tract cancer (esophageal, gastric, pancreatic and liver cancer). When planning the optimal therapy in patients with upper gastrointestinal malignancies it is essential to know the exact lymph node stage. Recently endoscopic sonoelastography(ES) has been added to conventional EUS examination and may provide complementary information to distinguish benign for malignant lymph nodes.

The N-stage relates to the treatment choice and the prognosis, and it is therefore of particular interest to know the interobserver agreement in operator dependent techniques. This study evaluate the interobserver agreement of EUS and ES evaluation og lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a lymph node more than 10mm in diameter (short axis) detected during the EUS examination

Exclusion Criteria:

* inadequate ES images were obtained by one of the observers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for EUS examination on the basis of a malignant indication.
Sampling Method: Non-Probability Sample
Enrollment: 74
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Larsen, MD, Principal Investigator
Locations (1):
- Centre for Surgical Ultrasound, Odense, Denmark